CLINICAL TRIAL: NCT06134362
Title: A Phase IIIB, Long-Term Follow-Up of CAB LA for Participants in HPTN 083 and HPTN 084 CAB PrEP Studies at Risk of HIV Acquisition
Brief Title: Long-term Follow-up of Long-acting Cabotegravir (CAB LA) for PrEP (Pre-exposure Prophylaxis) in Participants at Risk of Acquiring HIV (Human Immunodeficiency Virus)
Acronym: PALISADE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 221163
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections
Keywords: HIV; Human Immunodeficiency Virus; CAB LA; Cabotegravir; Apretude; PrEP; HPTN 083; HPTN 084; DAIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — cabotegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAB LA 600 mg (Q8W) (Experimental): All enrolled participants have previously received CAB LA as part of the HPTN 083 and HPTN 084 parent studies or their sub-studies. Participants will continue receiving CAB LA 600 mg via gluteal intramuscular (IM) injection.
  Interventions: Drug: CAB LA

INTERVENTIONS:
Drug: CAB LA — Participants will receive CAB LA 600 mg via gluteal IM injection, once every 8 weeks (Q8W).
  Other Names: Apretude; CAB LA for PrEP

SUMMARY:
The purpose of this study is long-term evaluation of long-acting injectable cabotegravir (CAB LA) for HIV pre-exposure prophylaxis (PrEP) in eligible participants who have completed DAIDS (Division of AIDS) sponsored studies HPTN 083 and HPTN 084 and associated sub-studies. Participants will continue receiving CAB LA and be followed for new HIV diagnosis, SAEs (serious adverse events), Grade 3 and Grade 4 ISRs (injection site reactions), and AEs (adverse events) leading to withdrawal.

ELIGIBILITY:
Inclusion criteria:

Type of participant

1. Participants must have recently completed or be currently enrolled and ongoing in one of the following studies on the CAB LA arm:

   * HPTN 083 open label extension
   * HPTN 084 open label extension (including pregnancy sub-study)

   Participants that completed study participation ≥3 months ago must be discussed with the Medical Monitor prior to enrolment.

   Participants who have prematurely withdrawn from prior CAB PrEP studies cannot enroll into this study.
2. Evidence of continued benefit (HIV negative and at risk) from CAB LA during participation in the parent study/sub-study.
3. Participants must have nonreactive HIV tests at Screening (rapid test, immunoassay [antigen/antibody] test and HIV-1 RNA results must all be available and nonreactive) and Day 1 (at least one of rapid test and immunoassay [antigen/antibody test] results must be available and nonreactive). Participants who have one or more reactive or positive HIV test result(s) will not be enrolled, even if subsequent confirmatory testing indicates they are not HIV-infected.

   Sex
4. Males and Females:

   All participants who are engaging in sexual activity should be counselled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom) and on the risk of acquiring HIV and other STIs.

   Females:

   Cisgender female participants who are of childbearing potential and who are engaging in sexual activity that could lead to pregnancy, must talk to the investigator about recommended contraception options. Contraception will be optional in this study. Condoms are recommended in addition, because their appropriate use is the only contraception method effective for preventing HIV-1 transmission.

   Pregnant participants from the HPTN 084 study are eligible to enroll into this study if they meet all eligibility criteria.

   Informed consent
5. Participant or caregiver/legal guardian is able and willing to provide signed informed consent as described in Protocol Section 11.1.5, which includes compliance with the requirements and restrictions listed in the consent form and in this protocol. Where applicable, participants must provide written assent.

Exclusion Criteria:

Concurrent conditions/medical history (includes liver function)

1. Participants who are currently enrolled in the eligible studies on the TDF/FTC arm are not eligible to enroll into this study. Participants receiving short-term oral TDF/FTC bridging may be enrolled following consultation with the Medical Monitor.
2. Previous premature discontinuation from IP in the parent study/sub-study.
3. ALT >5 × ULN; or ALT>3 × ULN and bilirubin >1.5 × ULN (with >35% direct bilirubin) in the screening liver chemistry test result.
4. Participants with known active hepatitis B infection (as indicated by a positive HBsAg and/or quantifiable HBV DNA). Participants negative for HBsAg but positive for anti-HBc and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.
5. Unstable liver disease (as defined by any of the following: presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice or cirrhosis), known biliary abnormalities (with the exception of hyperbilirubinemia or jaundice due to Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator).
6. Known history of cirrhosis with or without viral hepatitis co-infection.
7. Participant is currently participating in or has participated in a study (other than the studies listed in Inclusion Criteria 1) with a compound or device that is not commercially available within 30 days prior to signing informed consent, unless permission from the Medical Monitor is granted.
8. Presence of or any history of allergy/sensitivity to the study drug or its components.
9. Inflammatory skin conditions that compromise the safety of IM injections, per the discretion of the investigator. Mild skin conditions may not be exclusionary at the discretion of the investigator or designee.
10. Participant has a gluteal implant, tattoo or other dermatological condition overlying the buttock region which in the opinion of the investigator or designee may interfere with the injection or interpretation of ISRs.
11. Coagulopathy (primary or iatrogenic) which would contraindicate IM injection. Concomitant medications
12. Participant is receiving any protocol-defined prohibited medication and is unwilling or unable to switch to an alternate medication.
13. Anticipated need for HCV therapy with interferon or any drugs that have potential for adverse drug: drug interactions with study treatment throughout the entire study period.

    Relevant habits
14. Participant is unlikely to adhere to the study procedures, keep appointments, or is planning to relocate during the study.
15. Any condition (i(including but not limited to substance use disorder) that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol.

    Other
16. Participant has in the last 14 days prior to screening presented with signs and symptoms, which, in the opinion of the investigator, are suggestive of acute HIV infection. Participants may only be enrolled if clinical suspicion of HIV is ruled out with non-reactive results using appropriate HIV tests as per Inclusion Criterion #3.
17. Participant is a ward of the state (e.g. child in care).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3508 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with new HIV infection | From Day 1 up to end of study (up to approximately [approx.] 3 years)
Number of participants with new HIV infection by characteristic | From Day 1 up to end of study (up to approx. 3 years)
  Relevant characteristics of new HIV infections will be assessed, including presence of viral resistance to CAB.

SECONDARY OUTCOMES:
Number of participants with serious adverse events (SAE) by severity | From Day 1 up to end of study (up to approx. 3 years)
  The severity scale is assessed as following: Grade 1 = mild symptoms causing no or minimal interference with usual social and functional activities with intervention not indicated. Grade 2 = moderate symptoms causing greater than minimal interference with usual social and functional activities with intervention indicated. Grade 3 = severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated. Grade 4 = potentially life-threatening symptoms causing inability to perform self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death.
Number of participants with Grade 3 and Grade 4 injection site reactions (ISRs) | From Day 1 up to end of study (up to approx. 3 years)
  ISRs may occur following intramuscular administration of CAB LA. Grade 3 refers to severe symptoms causing inability to perform usual social & functional activities with intervention or hospitalization indicated. Grade 4 refers to potentially life-threatening symptoms causing inability to perform basic self-care functions with intervention indicated to prevent permanent impairment, persistent disability or death.
Number of participants with any clinical or laboratory AE leading to discontinuation of CAB LA, by severity | From Day 1 up to end of study (up to approx. 3 years)
  Any clinical or laboratory AE that leads the participant to permanently discontinue CAB LA will be assessed. The severity scale is assessed as following: Grade 1 = mild symptoms causing no or minimal interference with usual social and functional activities with intervention not indicated. Grade 2 = moderate symptoms causing greater than minimal interference with usual social and functional activities with intervention indicated. Grade 3 = severe symptoms causing inability to perform usual social and functional activities with intervention or hospitalization indicated. Grade 4 = potentially life-threatening symptoms causing inability to perform self-care functions with intervention indicated to prevent permanent impairment, persistent disability, or death.

CONTACTS AND LOCATIONS:
Locations (24):
- Argentina (2):
  - GSK Investigational Site, Almagro
  - GSK Investigational Site, Buenos Aires
- GSK Investigational Site, Francistown, Botswana
- Brazil (3):
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo
- GSK Investigational Site, Mbabane, Eswatini
- GSK Investigational Site, Kisumu, Kenya
- Malawi (2):
  - GSK Investigational Site, Blantyre
  - GSK Investigational Site, Lilongwe
- Peru (2):
  - GSK Investigational Site, Lima
  - GSK Investigational Site, Piura
- South Africa (6):
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, City of Cape Town
  - GSK Investigational Site, City of Johannesburg
  - GSK Investigational Site, Durban
  - GSK Investigational Site, Isipingo
  - GSK Investigational Site, Sol Plaatjie
- Thailand (2):
  - GSK Investigational Site, Chiang Mai, Chiang Mai
  - GSK Investigational Site, Pathum Wan
- Uganda (2):
  - GSK Investigational Site, Entebbe
  - GSK Investigational Site, Kampala
- Zimbabwe (2):
  - GSK Investigational Site, Chitungwiza
  - GSK Investigational Site, Harare

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf